CLINICAL TRIAL: NCT04359043
Title: The Acceptability and Feasibility of an Adaptation of The Mediational Intervention for Sensitizing Caregivers for Community Based Organizations in a Sample of South African HIV/AIDS Orphans
Brief Title: MISC-CBO in Children Affected by HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of the Free State (Unknown); Michigan State University (Other); Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Carla Sharp, Professor, University of Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15598-02
Record Dates: First submitted 2020-04-09; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: HIV Affected Children (Single and/or Double Orphans)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This was a quasi-experimental study with two treatment arms: intervention vs. TAU. Subjects were not randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediational Intervention for Sensitizing Caregivers (Experimental): Half of the child participants and the careworkers in the Community-based Organization taking care of them, received the Mediational Intervention for Sensitizing Caregivers.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC)
- Treatment as Usual (Other): The other half of child participants and the careworkers in the Community-based Organization taking care of them, received Treatment as Usual which consists of the usual services delivered to children at the CBO: food, help with homework, registrations for birth certificates.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC) — MISC is an intervention that focuses on increasing the caregiving capacity of the caregiver by enhancing a set of emotional and cognitive components that collectively, sensitizes the caregiver to the emotional and cognitive needs of the child.
  Arms: Mediational Intervention for Sensitizing Caregivers
Behavioral: Treatment as Usual — Treatment as Usual was delivered by community-based organization caseworkers. It consists of a nutritional curriculum of the same dosage and time commitment as the experimental condition, but with no caregiving component.
  Arms: Treatment as Usual

SUMMARY:
Currently, 12 million children in Sub-Saharan Africa and 1.9 million children in South Africa (SA) are orphaned by HIV/AIDS. Research addressing what can be done to support these children has been limited, clustered and of variable quality. Our prior work showed that an important support structure for care of HIV affected children (orphans) in SA is through Community Based Organizations (CBOs). Currently, no evidence-based CBO intervention exist. CBO careworkers report low efficacy in addressing the mental health and cognitive developmental needs of children. There is therefore a critical need to empower frontline CBO careworkers to be trained in addressing the mental health and cognitive developmental needs of orphans. The Mediational Intervention for Sensitizing Caregivers (MISC) used in our previous work with parents in Uganda holds promise. The objective in this application is to use a mixed methods approach (observations, focus groups, questionnaires) to test the acceptability and feasibility of adapting MISC to be used by CBO careworkers instead of parents (MISC-CBO), and to assess preliminary outcomes. Guided by the Mathews and Hudson's framework for evaluating caregiver-child training programs, our approach will consist of three phases: Adapt, Process evaluation, Outcome evaluation. In Phase 1 (Adapt, Year 1) we will conduct formative research (qualitative interviews and focus groups) with community stakeholders, a Community Advisory Board and children to ascertain feasibility and acceptability of MISC-CBO in the SA cultural context with 7-11 year old AIDS orphans. In Phase 2 (Implementation and process evaluation, Year 2) we will recruit 80 AIDS orphans through 4 CBOs (20 children and 4 careworkers from each CBO). Two CBOs will be allocated to MISC-CBO and 2 will be allocated to treatment as usual (TAU of comparable contact hours). One year of bi-weekly (every 2 weeks) intervention sessions will be conducted. Process evaluation will include individual interviews, observations, focus groups and questionnaire-based assessment of MISC-CBO feasibility, adherence and fidelity. In Phase 3 (Outcomes assessment, Years 2 & 3) the effects of MISC-CBO to promote mental health and cognitive development through the mechanism of improved quality of caregiving by CBO careworkers will be assessed through mental health and cognitive assessments at baseline (beginning of Year 2), 6, 12 and 18 months compared to TAU in the children and careworkers recruited in Phase 2. At the end of this formative RO1 that transforms a parent intervention into a CBO careworker intervention, we will have established the foundational assessments and intervention to apply for an RO1 to evaluate a randomized controlled trial designed to fully test the efficacy of MISC-CBO during the critical developmental window of at-risk HIV affected children aging into adolescence. This project will make possible the only culture-appropriate and sustainable evidence-based CBO intervention that can be readily and effectively implemented globally in low-resource settings with children generally at risk from disease, malnutrition and neglect.

DETAILED DESCRIPTION:
Currently, 12 million children in Sub-Saharan Africa and 1.9 million children in South Africa (SA) are orphaned by HIV/AIDS1. Research addressing what can be done to support these children has been limited, clustered and of variable quality2. Our prior work in SA (PI: Sharp; R01 MH078757) showed that an important care support structure for orphans is through Community Based Organizations (CBOs). Currently, no evidence-based CBO interventions exist. Moreover, CBO careworkers report a desire to learn how to address the mental health and cognitive developmental needs of children3. There is a critical need to empower frontline CBO careworkers to be trained in how to respond to the mental health and cognitive developmental needs of orphans. The Mediational Intervention for Sensitizing Caregivers (MISC)4-6 used in our previous work (PI: Boivin; R34 MH082663; RO1 HD070723) with parents in Uganda holds promise. The objective of this application is to use a mixed methods approach to test the acceptability and feasibility of adapting MISC for CBOs (MISC-CBO), and to assess preliminary outcomes. Guided by the Mathews and Hudson's framework for evaluating caregiver-child training programs7, our approach will consist of three phases: Adapt, Process Evaluation, Outcome Evaluation. Our central hypothesis is that feasibility and acceptability of MISC-CBO will be established and that positive preliminary outcomes will be demonstrated.

Aim 1: Adapt MISC to establish acceptability of MISC-CBO (Yr 1). We will conduct formative research (qualitative interviews and focus groups) with community stakeholders, a Community Advisory Board (CAB) and children to ascertain feasibility and acceptability of MISC-CBO with 7-11 year olds affected by HIV/AIDS in SA. Hyp1: Formative work will result in an adaptation of MISC that is deemed acceptable.

Aim 2: Implementation and process evaluation of MISC-CBO to establish feasibility, adherence and fidelity (Yr 2). We will recruit N = 80 HIV/AIDS orphans through 4 CBOs (i.e. 20 children, 4 careworkers and CBO director from each CBO). Two CBOs will be allocated to MISC-CBO while the other 2 will be allocated to treatment as usual (TAU of comparable contact hours). After initial training, one year of bi-weekly (every 2 weeks) intervention sessions of MISC-CBO and TAU will be conducted. Process evaluation will include individual interviews, observations, focus groups and questionnaire-based assessment of feasibility of the intervention perceived by CBO careworkers, directors and children themselves. MISC-CBO adherence and fidelity will be assessed. Hyp2: CBO careworkers and directors will readily and reliably participate in bi-weekly MISC-CBO training and evaluation. Hyp3: Qualitative interviews will show that CBO careworkers and directors support the goals and affordability of MISC-CBO. Hyp4: Video footage and questionnaire data will show fidelity to MISC-CBO in terms of content and caregiving adherence.

Aim 3: Outcomes evaluation of MISC-CBO (Yrs 2 & 3). The effects of MISC-CBO on mental health and cognitive development through the mechanism of improved quality of CBO caregiving will be assessed through assessments at baseline (the beginning of Yr 2), 6, 12 and 18 months compared to TAU in the children and careworkers recruited in Aim 2. Hyp5: MISC-CBO careworkers will have significantly more positive interactions with study children compared with TAU careworkers. Hyp6: Children in MISC-CBO will show reduction in symptoms of emotional and behavior problems and increased behaviors indicative of positive emotional outcomes as determined by observations and questionnaire data. Hyp7: Children in MISC-CBO's cognitive ability tests scores will improve. Hyp8: The cognitive and mental health gains for children will be statistically mediated by improved caregiving quality and increased knowledge of MISC principles in MISC-CBO workers.

Overall impact. This is a small-scale, developmental 3-year RO1 that builds on our established US-SA-NIH partnerships (Sharp, Marais, Skinner, Serekoane) to develop an expanded research team (adding MISC experts Boivin and Klein), and create a CAB to assist in the adaptation of MISC for CBOs. Our proposed research is in line with the NIH priorities as well as UNICEF's goal of strengthening the capacities of communities, and fits with our long-term research goal to address the mental health needs of HIV/AIDS affected children. At the end of this formative study, we will have established the foundational assessments and intervention to apply for an RO1 to evaluate a randomized controlled trial designed to fully test the efficacy of MISC-CBO during the critical developmental window of at-risk HIV affected children aging into adolescence. This project will make possible the only culture-appropriate and sustainable evidence-based CBO intervention that can be readily and effectively implemented globally in low-resource settings with children generally at risk from disease, malnutrition and neglect.

ELIGIBILITY:
Inclusion Criteria:

* orphaned (UNICEF criterion of one or both parents deceased from AIDS)
* HIV/AIDS affected child as determined by verbal autopsy measure to determine cause of death of biological parent(s)
* 7-11 year old
* resident in the CBO catchment area
* principle home caregiver of the child should be able to participate in baseline and follow-up assessments

Exclusion Criteria:

* medical history of serious birth complications
* severe malnutrition, bacterial meningitis
* encephalitis
* cerebral malaria
* known brain injury or disorder requiring hospitalization
* continued evidence of seizure or other neurological disability
* HIV infection

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Strengths and Difficulties Questionnaire (SDQ) Total Score as index of improvement in overall mental health in children | baseline, 6 months follow-up, 12 months follow-up
  The Strengths and Difficulties Questionnaire (Goodman, 2001) is a well validated measure of mental health in children. While the measure covers several domains of emotional-behavioral psychiatric symptoms (anxiety, depression, conduct problems, peer problems and prosocial behavior), it is most often summed to derive a total score to index overall level of mental health problems in children. The use of this measure in this way has been validated in a Sesotho speaking population of children where it was shown that the total score provides a good index of mental health problems in HIV/AIDS affected children (Sharp et al., 2014). This measure has also been shown to be sensitive to change and therefore serves as a good outcome measure to assess overall improvement in mental health as a function of our behavioral intervention.
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to Focus the child. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The cognitive components include the following subscale: Focusing, Providing meaning, Expanding, Regulating, and Rewarding. The Focusing subscale assesses the caregiver's capacity to focus the child's attention on a topic or object. It is the first step in providing a mediational learning experience for a child and one of the outcomes that the MISC intervention targets. The OMI tallies each instance when Focusing occurs during a 7-minute video-taped interaction. This is the unit of measurement for the OMI Focusing outcome that will be assessed here. An example of a behavior that is coded as Focusing is: "Look here!".
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to Provide meaning to the child's subjective experience. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The cognitive components include the following subscale: Focusing, Providing meaning, Expanding, Regulating, and Rewarding. The Provision of meaning subscale assesses the caregiver's capacity to describe the subjective experience of the child. The OMI tallies each instance when Provision of meaning occurs during a 7-minute video-taped interaction. This is the unit of measurement for the OMI Provision of meaning outcome that will be assessed here. An example of a behavior that is coded as Provision of meaning is: "This is a butterly!"
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to Expand the child's learning. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The cognitive components include the following subscale: Focusing, Providing meaning, Expanding, Regulating, and Rewarding. The Expanding subscale assesses the caregiver's capacity to expand the child's learning around the topic under discussion. The OMI tallies each instance when Expanding occurs during a 7-minute video-taped interaction. This is the unit of measurement for the OMI Expanding outcome that will be assessed here. An example of a behavior that is coded as Expanding is: "Butterflies are important for pollination of flowers".
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to Regulate the child. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The cognitive components include the following subscale: Focusing, Providing meaning, Expanding, Regulating, and Rewarding. The Regulating subscale assesses the caregiver's capacity to regulate the child's learning around the topic under discussion. The OMI tallies each instance when Regulating occurs during a 7-minute video-taped interaction. This is the unit of measurement for the OMI Regulating outcome that will be assessed here. An example of a behavior that is coded as Regulating is: "To build the tower, we must first put down the big block; then you can put down the small block".
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to Reward the child. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The cognitive components include the following subscale: Focusing, Providing meaning, Expanding, Regulating, and Rewarding. The Rewarding subscale assesses the caregiver's capacity to reward the child during interaction. The OMI tallies each instance when Rewarding occurs during a 7-minute video-taped interaction. This is the unit of measurement for the OMI Rewarding outcome that will be assessed here. An example of a behavior that is coded as Rewarding is: "Well done. You were very careful in placing the blocks on top of each other so that they don't fall down".
Change in Observed Mediational Interactions (OMI; Klein, 1996) score in the caregiver's capacity to utilize affective components. | baseline, 6 months follow-up, 12 months follow-up
  The OMI is an observational measure of caregiver-child interactions. Interactions between caregiver and child are video-recorded and the components of a mediated learning experience is then coded using the OMI coding manual. Mediated learning components include two sets of measurements: cognitive and affective components. The affective components are several behaviors that the observer codes, each on a 5 point scale. These include smiling, synchrony, turntaking, touching, validating, and positive affect. The scores on each of these behaviors are then totaled to provide a total score on affective components observed during the 7-minute videotaped interaction.
Change in the Kaufman Brief Intelligence Test (KBIT) overall IQ composite | baseline, 6 months follow-up, 12 months follow-up
  The Kaufman Brief Intelligence Test (KBIT) (Kaufman & Kaufman, 2004) is a brief, individually administered measure of verbal (vocabulary subtest) and non verbal (Matrices subtest) intelligence. It can be used with those aged 4-90 years old and takes between 15-30 minutes to administer. The KBIT-2 generates three scores: Verbal, Non Verbal and an overall IQ composite. Theoretically the verbal subtests measure crystallised ability and the non verbal subtests measure fluid reasoning. The KBIT has been used successfully in South Africa (Ogunlade, A.O., et al.2011) and neuropsychologist and Co-Investigator Boivin has been using it in Johannesburg in yet unpublished work with the relevant population for the current research. The overall IQ composite will be used to assess change in cognitive outcomes as a function of the MISC intervention.
Change in Behavior Rating Inventory of Executive Function (BRIEF) Global Executive Composite score to assess change in executive functions as a function of the intervention. | baseline, 6 months follow-up, 12 months follow-up
  The Behavior Rating Inventory of Executive Function (BRIEF-) (Gioia et al., 2003) is useful for evaluating and planning treatment strategies for a wide spectrum of developmental and acquired neurological conditions, including learning disabilities, low birth weight, ADHD, Tourette's disorder, traumatic brain injury, and autism. These scales include the behavior/cognitive functions of Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials, and Monitor. Given this focus, the BRIEF will complement, rather than overlap with the Strengths and Difficulties Questionnaire used for more general mental health problems. The eight non-overlapping clinical scales form two broader indexes: Behavior Regulation (three scales) and Metacognition (five scales). A Global Executive Composite score is also produced. This is our principal outcome measure from this assessment. A Sesotho version of the measure was obtained through the publisher.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Development Support Center, UFS, Bloemfontein, Free State, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
Not clear yet. Needs discussion with IRB given the vulnerable population.